CLINICAL TRIAL: NCT04129164
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Proof of Concept Study to Evaluate the Efficacy and Safety of VIB4920 in Subjects With Sjögren's Syndrome (SS)
Brief Title: A Study to Evaluate the Efficacy and Safety of VIB4920 in Participants With Sjögren's Syndrome
Acronym: SS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIB4920.P2.S2; 2019-002713-19 (EudraCT Number)
Record Dates: First submitted 2019-10-02; First posted 2019-10-16 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Sjögren's Syndrome
Keywords: Sjögren's Syndrome; SS; VIB4920; MEDI4920
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VIB4920 Dose 1 in Population 1 (Experimental): Participants in population 1 will receive IV VIB4920 Dose 1 in Stage I and placebo matched to VIB4920 in Stage II.
  Interventions: Drug: VIB4920; Drug: Placebo
- Placebo in Population 1 (Placebo Comparator): Participants in population 1 will receive IV placebo matched to VIB4920 in Stage I and IV VIB4920 Dose 1 in Stage II.
  Interventions: Drug: VIB4920; Drug: Placebo
- VIB4920 Dose 1 in Population 2 (Experimental): Participants in population 2 will receive IV VIB4920 Dose 1 in Stage I and placebo matched to VIB4920 in Stage II.
  Interventions: Drug: VIB4920; Drug: Placebo
- Placebo in Population 2 (Placebo Comparator): Participants in population 2 will receive IV placebo matched to VIB4920 in Stage I and IV VIB4920 Dose 1 in Stage II.
  Interventions: Drug: VIB4920; Drug: Placebo

INTERVENTIONS:
Drug: VIB4920 — Intravenous Dose 1.
  Other Names: Dazodalibep
Drug: Placebo — Intravenous dose matched to VIB4920.

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and tolerability of VIB4920 (formerly MEDI4920) in adult participants with Sjögren's Syndrome (SS).

DETAILED DESCRIPTION:
The study will enrol 2 SS populations: Population 1 will include participants with moderate to high systemic disease activity defined by European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI) >= 5; Population 2 will include participants with moderate to severe subjective symptoms defined by EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) score >= 5 and residual stimulated salivary flow but with mild systemic disease activity defined by ESSDAI score < 5. This study will include 3 periods: screening (4 weeks), treatment period (40 Weeks) and follow-up period (12 weeks). In the treatment period, participants from each of the populations will be randomized at 1:1 ratio to receive intravenous (IV) dose of VIB4920 or placebo (Stage I). After completion of Stage I, participants randomized to VIB4920 in Stage I will receive placebo and participants randomized to placebo in Stage I will receive VIB4920 (Stage II). Participants who had study drug discontinuation will not be eligible for treatment during Stage II. All participants will be followed for at least 12 weeks after their last dose of study drug administration.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SS by meeting the 2016 American College of Rheumatology (ACR)/EULAR Classification Criteria.
* Residual salivary gland function as defined by whole stimulated salivary flow > 0.1 mL/min (only for Population 2).
* Have an ESSDAI score of >= 5 at screening; (not including the peripheral nervous system, central nervous system, and pulmonary domains) (only for Population 1).
* Have an ESSPRI score of >= 5 at screening (only for Population 2).
* Have an ESSDAI score of < 5 at screening (only for Population 2).
* Positive for either anti-Ro autoantibodies or rheumatoid factor, or both at screening.
* Male and female participants who agree to follow protocol defined contraceptive methods.
* No active or untreated latent tuberculosis (TB).

Exclusion Criteria:

* Medical history of confirmed deep venous thrombosis or arterial thromboembolism within 2 years of signing the informed consent form (ICF).
* Risk factors for venous thromboembolism or arterial thrombosis, prothrombotic status.
* Concomitant polymyositis or dermatomyositis or systemic sclerosis.
* Active malignancy or history of malignancy, except in situ carcinoma of the cervix and cutaneous basal cell carcinoma.
* Hepatitis B, hepatitis C, or human immunodeficiency virus infection.
* More than one episode of herpes zoster and/or an opportunistic infection in the last 12 months.
* Active viral, bacterial, or other infections or history of more than 2 infections requiring intravenous antibiotics within 12 months prior to signing the ICF.
* Participants with corona virus disease 2019 (COVID-19) infection or who, in the judgment of the investigator, are at unacceptable risk of COVID-19 or its complications.
* A documented positive severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) test within 2 weeks prior to randomization.
* Received live (attenuated) vaccine within the 4 weeks prior to ICF signature.
* Treated with any biologic B-cell-depleting therapy within 12 months or other B-cell targeting therapy < 3 months before randomization.
* Injectable corticosteroids (including intraarticular) or treatment with > 10 mg/day dose oral prednisone or equivalent within 6 weeks prior to randomization (only for Population 1).
* Treated with systemic corticosteroids for indications other than SS, rheumatoid arthritis (RA), and systemic lupus erythematosus (SLE) for more than a total of 2 weeks within 24 weeks prior to screening visit (only for Population 1).
* Received previous treatment with anti-CD40L compounds at any time before screening.
* Pregnant or lactating or planning to get pregnant during the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (56):
- United States (15):
  - Research Site, Fullerton, California
  - Research site, Upland, California
  - Research Site, Lawrenceville, Georgia
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Wheaton, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research site, Duncansville, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research site, Dallas, Texas
  - Research Site, Houston, Texas
- Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina
- France (5):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Grenoble
  - Research Site, Paris
  - Research Site, Strasbourg
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
- India (6):
  - Research Site, Secunderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Pune, Maharshtra
  - Research Site, Bhubaneswar, Odisha
  - Research Site, Chennai, Tamil Nadu
- Italy (6):
  - Research Site, Milan, Lambardia
  - Research Site, Rome, Lazio
  - Research Site, Brescia, Province Of Brescia
  - Research Site, Perugia, Umbria
  - Research Site, Pisa
  - Research Site, Udine
- Mexico (3):
  - Research Site, Saltillo, Coahuila
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City
- Peru (2):
  - Research Site, Lima, San Martin de Porres
  - Research Site, Lima
- Poland (8):
  - Research Site, Elblag, Elblag
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Siedlce
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- South Korea (3):
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Incheon, Republic of Korea
  - Research Site, Seoul, Republic of Korea
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
- United Kingdom (2):
  - Research Site, Newcastle upon Tyne
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St Clair EW, Baer AN, Ng WF, Noaiseh G, Baldini C, Tarrant TK, Papas A, Devauchelle-Pensec V, Wang L, Xu W, Pham TH, Sikora K, Rees WA, Alevizos I. CD40 ligand antagonist dazodalibep in Sjogren's disease: a randomized, double-blinded, placebo-controlled, phase 2 trial. Nat Med. 2024 Jun;30(6):1583-1592. doi: 10.1038/s41591-024-03009-3. Epub 2024 Jun 5. PMID 38839899
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 70 international sites between November 2019 and March 2023.
Pre-assignment Details: Eligibility for Sjögren's syndrome (SS) was assessed using the 2016 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria. Participants were then randomized into a double-blind treatment period and categorized into two populations based on the severity of systemic disease activity and symptoms.
Groups:
- Population 1: Placebo/VIB4920: Participants with SS characterized by moderate to severe systemic disease activity (defined by an ESSDAI score of ≥ 5), were randomized to receive a placebo in Stage I, followed by VIB4920 in Stage II.
- Population 1: VIB4920/Placebo: Participants with SS characterized by moderate to severe systemic disease activity (defined by a ESSDAI score of ≥ 5), were randomized to receive multiple doses of VIB4920 in Stage I, followed by a placebo in Stage II.
- Population 2: Placebo/VIB4920: Participants with SS characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), were randomized to receive a placebo in Stage I, followed by VIB4920 in Stage II.
- Population 2: VIB4920/Placebo: Participants with SS, characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), were randomized to receive multiple doses of VIB4920 in Stage I, followed by a placebo in Stage II.
Period: Overall Study
Arm/Group | Population 1: Placebo/VIB4920 | Population 1: VIB4920/Placebo | Population 2: Placebo/VIB4920 | Population 2: VIB4920/Placebo
Started | 38 | 36 | 55 | 54
Completed Stage I | 37 | 34 | 52 | 49
Completed | 35 | 32 | 47 | 47
Not Completed | 3 | 4 | 8 | 7
Not completed — Non-compliance with procedures | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 4 | 6
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): included all randomized participants who received any dose of investigational product, analyzed according to the randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Population 1: Placebo/VIB4920 | Population 1: VIB4920/Placebo | Population 2: Placebo/VIB4920 | Population 2: VIB4920/Placebo | Total
Number analyzed (Participants) | 38 | 36 | 55 | 54 | 183
Age, Customized [Number; unit: participants]
  18-85 years | 38 | 36 | 55 | 54 | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 50 | 53 | 176
  Male | 0 | 1 | 5 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 23 | 22 | 61
  Not Hispanic or Latino | 30 | 28 | 32 | 32 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 11 | 9 | 25
  Asian | 0 | 2 | 5 | 11 | 18
  Black or African American | 1 | 3 | 3 | 4 | 11
  White | 34 | 26 | 31 | 23 | 114
  Other | 2 | 1 | 5 | 7 | 15
Population 1: Baseline ESSDAI Total Score [Mean (Standard Deviation); unit: score on scale] — The ESSDAI is a systemic disease activity index for SS, assessing 12 domains (Constitutional, Salivary Glands, Lungs, Kidneys, Musculoskeletal, Peripheral Nervous System, Central Nervous System, Vascular, Gastrointestinal, Hematological, Ocular, and Extraglandular Manifestations). The final score is calculated as the sum of all weighted domain scores. The theoretical range is 0 to 123, with lower scores indicating less disease activity. Population: The baseline ESSDAI total score for Population 1 is reported to support the primary outcome measure and is not collected for the overall study population.
  score on scale
    number analyzed (Participants) | 38 | 36 | 0 | 0 | 74
    (all) | 10.1 (4.1) | 11.4 (4.5) |  |  | 10.7 (4.3)
Population 2: Baseline ESSPRI Total Score [Mean (Standard Deviation); unit: score on a scale] — The ESSPRI is a self-assessment tool for evaluating symptoms of dryness, fatigue, and pain (articular and/or muscular) in SS. Participants rate each of the three domains on a 0-10 numerical scale (0 = no; 10 maximal imaginable severity). All domains are equally weighted, and the total score is the mean of the three domain scores. The maximum total score for the ESSPRI assessment is 10. Population: The baseline ESSPRI total score for Population 2 is reported to support the primary outcome measure and is not collected for the overall study population, including Population 1.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 55 | 54 | 109
    (all) |  |  | 6.8 (1.2) | 7.1 (1.6) | 6.9 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Population 1: Change From Baseline in ESSDAI at Day 169
Description: The ESSDAI is a systemic disease activity index for SS, assessing 12 domains (Constitutional, Salivary Glands, Lungs, Kidneys, Musculoskeletal, Peripheral Nervous System, Central Nervous System, Vascular, Gastrointestinal, Hematological, Ocular, and Extraglandular Manifestations). Each domain is graded for activity (0 = no activity to 3 = high activity) and weighted (1 for Biological to 6 for Muscular) based on its clinical significance, with the final score calculated as the sum of all weighted domain scores. The theoretical range is 0 to 123, with disease activity categorized as low (<5), moderate (5-13), and high (≥14). A positive change form baseline represents an increase in symptoms.
Time Frame: Baseline and Day 169
Population: FAS: included all randomized participants who received any dose of investigational product, analyzed according to the randomized treatment, and had available data at the specified time points.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Groups:
- Population 1: Placebo: Participants with SS characterized by moderate to severe systemic disease activity (defined by an ESSDAI score of ≥ 5), were randomized to receive a placebo in Stage I.
- Population 1: VIB4920: Participants with SS characterized by moderate to severe systemic disease activity (defined by a ESSDAI score of ≥ 5), were randomized to receive multiple doses of VIB4920 in Stage I.
Arm/Group | Population 1: Placebo | Population 1: VIB4920
Number analyzed (Participants) | 36 | 33
Score on scale | -4.1 (0.6) | -6.3 (0.6)

2. Primary Outcome: Population 2: Change From Baseline in ESSPRI at Day 169
Description: The ESSPRI is a self-assessment tool for evaluating symptoms of dryness, fatigue, and pain (articular and/or muscular) in SS. Participants rate each of the three domains on a 0-10 numerical scale (0 = no; 10 maximal imaginable severity). All domains are equally weighted, and the total score is the mean of the three domain scores. The maximum total score for the ESSPRI assessment is 10. A positive change form baseline represents an increase in symptoms.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Groups:
- Population 2: Placebo: Participants with SS characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), were randomized to receive a placebo in Stage I.
- Population 2: VIB4920: Participants with SS, characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), were randomized to receive multiple doses of VIB4920 in Stage I.
Arm/Group | Population 2: Placebo | Population 2: VIB4920
Number analyzed (Participants) | 53 | 51
Score on scale | -0.53 (0.23) | -1.80 (0.23)

3. Secondary Outcome: Population 1: Change From Baseline in ESSPRI at Day 169
Description: The ESSPRI is a self-assessment tool for evaluating symptoms of dryness, fatigue, and pain (articular and/or muscular) in SS. Participants rate each of the three domains on a 0-10 numerical scale (0 = no; 10 maximal imaginable severity). All domains are equally weighted, and the total score is the mean of the three domain scores. The maximum total score for the ESSPRI assessment is 10. A positive change from baseline represents an increase in symptoms.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Population 1: Placebo | Population 1: VIB4920
Number analyzed (Participants) | 36 | 33
Score on scale | -1.12 (0.29) | -1.80 (0.31)

4. Secondary Outcome: Population 1: Number of Participants Who Achieved ESSDAI[3] and ESSDAI[4] Response at Day 169
Description: The ESSDAI is a systemic disease activity index for primary Sjögren's syndrome, assessing 12 domains (e.g., cutaneous, renal, CNS, and biological). Each domain is graded for activity (0 = no activity to 3 = high activity) and weighted (1 for Biological to 6 for Muscular) based on its clinical significance, with the final score calculated as the sum of all weighted domain scores. The theoretical range is 0 to 123, with disease activity categorized as low (<5), moderate (5-13), and high (≥14). A positive change from baseline represents an increase in symptoms.
  ESSEDAI[3] and [4] responses were defined as a decrease of at least 3 or 4 points respectively in the ESSDAI score from the baseline value, measured at Day 169.
Time Frame: Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Population 1: Placebo | Population 1: VIB4920
Number analyzed (Participants) | 37 | 36
Participants
  ESSDAI[3] Day 169 | 22 | 26
  ESSDAI[4] Day 169 | 18 | 24

5. Secondary Outcome: Change From Baseline in The Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Day 169
Description: The FACIT-Fatigue is a 13-item patient-reported questionnaire designed to assess the impact of fatigue on quality of life (QoL). Responses are scored from 0 (Not at all) to 4 (Very Much). The total score is the sum of all responses, ranging from 0 to 52, with higher scores indicating better QoL. A positive change from baseline represents an increase in QoL.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Population 1: Placebo | Population 1: VIB4920 | Population 2: Placebo | Population 2: VIB4920
Number analyzed (Participants) | 36 | 33 | 52 | 51
Score on scale | 5.8 (1.6) | 8.1 (1.6) | 2.8 (1.4) | 8.1 (1.4)

6. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) at Day 169
Description: The OSDI is a validated tool for assessing vision-related function and dry eye disease severity (normal, mild, moderate, severe). It consists of 12 questions, with responses ranging from 0 (None of the time) to 4 (All of the time). Scores range from 0 to 100, as it is calculated by transforming the raw responses from the 12 questions into a standardized 0-100 scale, with higher scores indicating greater disability. A positive change from baseline indicates a worsening vision-related function.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Population 1: Placebo | Population 1: VIB4920 | Population 2: Placebo | Population 2: VIB4920
Number analyzed (Participants) | 35 | 31 | 50 | 51
Score on scale | -14.02 (3.06) | -16.00 (3.22) | -8.52 (2.94) | -13.95 (2.95)

7. Secondary Outcome: Patient Global Impression of Severity (PGIS) Score at Day 169
Description: The PGIS is a single-item measure that captures a patient's perception of overall symptom severity over the past week, using a 5-point categorical response scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe), with higher scores indicating greater symptom severity. Positive change from baseline values indicate worsening of symptoms severity.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Population 1: Placebo | Population 1: VIB4920 | Population 2: Placebo | Population 2: VIB4920
Number analyzed (Participants) | 36 | 33 | 52 | 51
Score on scale | -0.5 (0.1) | -0.6 (0.1) | -0.4 (0.1) | -0.6 (0.1)

8. Secondary Outcome: Population 2: Number of Participants Who Achieved ESSPRI Response at Day 169
Description: The ESSPRI is a self-assessment tool for evaluating symptoms of dryness, fatigue, and pain (articular and/or muscular) in SS. Participants rate each of the three domains on a 0-10 numerical scale (0 = no; 10 maximal imaginable severity). All domains are equally weighted, and the total score is the mean of the three domain scores. The maximum total score for the ESSPRI assessment is 10. A positive change form baseline represents an increase in symptoms. Participants achieving an ESSPRI response were defined as at least a 1 point or 15% reduction from baseline in ESSPRI score at Day 169 without premature discontinuation from the study and without receiving rescue medications.
Time Frame: Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Population 2: Placebo | Population 2: VIB4920
Number analyzed (Participants) | 55 | 54
Participants | 18 | 36

9. Secondary Outcome: Number of Participants Who Experience Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) referred to any untoward medical occurrence in a clinical study participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received the study treatment. Clinically significant changes in vital signs, electrocardiograms, and laboratory tests recorded after treatment administration were documented as TEAEs. Serious TEAEs (SAEs) were untoward medical occurrences after the first dose, irrespective of a causal link to the study treatment, that led to death, were life-threatening, required hospitalization or its prolongation, caused significant disability, resulted in congenital anomalies, or were considered other medically important events. AEs were graded (Grade 3: severe; Grade 4: life-threatening; Grade 5: death) using the Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Up to approximately 365 days
Population: Safety Analysis Set: included all participants who received any dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Population 1: Placebo/VIB4920 | Population 1: VIB4920/Placebo | Population 2: Placebo/VIB4920 | Population 2: VIB4920/Placebo
Number analyzed (Participants) | 38 | 36 | 55 | 54
Participants
  Stage 1 TEAEs | 23 | 28 | 38 | 37
  Stage 1 SAEs | 0 | 1 | 1 | 3
  Stage 1 Grade ≥ 3 | 0 | 2 | 1 | 2
  Stage 1 Fatal AEs | 0 | 1 | 0 | 0
  Stage 2 TEAEs: number analyzed (Participants) | 37 | 34 | 52 | 49
  Stage 2 TEAEs | 28 | 25 | 34 | 32
  Stage 2 SAEs: number analyzed (Participants) | 37 | 34 | 52 | 49
  Stage 2 SAEs | 1 | 3 | 1 | 2
  Stage 2 Grade ≥ 3: number analyzed (Participants) | 37 | 34 | 52 | 49
  Stage 2 Grade ≥ 3 | 0 | 2 | 0 | 3
  Stage 2 Fatal AEs: number analyzed (Participants) | 37 | 34 | 52 | 49
  Stage 2 Fatal AEs | 0 | 0 | 0 | 0

10. Secondary Outcome: Serum Concentration of VIB4920
Description: Blood samples were collected at the specified time points.
Time Frame: Day 1 pre-dose, Day 1 post-dose, Day 15, Day 29, Day 57, Day 85, Day 113, Day 141 pre-dose, Day 141 post-dose, Day 169 pre-dose, Day 169 post-dose, Day 197, Day 225, Day 253, Day 281, Day 309, Day 365
Population: Pharmacokinetic (PK) Analysis Set: included all participants who received investigational product and had at least one quantifiable plasma PK observation post-first dose.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Population 1: Placebo/VIB4920 | Population 1: VIB4920/Placebo | Population 2: Placebo/VIB4920 | Population 2: VIB4920/Placebo
Number analyzed (Participants) | 37 | 36 | 52 | 54
mg/L
  Day 1 pre-dose: number analyzed (Participants) | 0 | 36 | 0 | 54
  Day 1 pre-dose |  | 0.002 (0.013) |  | 0.002 (0.013)
  Day 1 post-dose: number analyzed (Participants) | 0 | 33 | 0 | 52
  Day 1 post-dose |  | 470.370 (111.047) |  | 496.984 (182.915)
  Day 15: number analyzed (Participants) | 0 | 35 | 0 | 51
  Day 15 |  | 97.058 (26.480) |  | 111.636 (56.244)
  Day 29: number analyzed (Participants) | 0 | 35 | 0 | 52
  Day 29 |  | 128.228 (31.805) |  | 141.365 (100.163)
  Day 57: number analyzed (Participants) | 0 | 34 | 0 | 51
  Day 57 |  | 62.363 (25.562) |  | 80.093 (64.358)
  Day 85: number analyzed (Participants) | 0 | 36 | 0 | 51
  Day 85 |  | 53.716 (21.300) |  | 68.812 (60.349)
  Day 113: number analyzed (Participants) | 0 | 31 | 0 | 50
  Day 113 |  | 52.796 (29.229) |  | 66.778 (59.558)
  Day 141 pre-dose: number analyzed (Participants) | 0 | 35 | 0 | 48
  Day 141 pre-dose |  | 49.318 (27.952) |  | 80.912 (125.684)
  Day 141 post-dose: number analyzed (Participants) | 1 | 33 | 1 | 47
  Day 141 post-dose | 0.577 (NA) — Standard deviation was not calculated as only one participant had PK observations. | 525.702 (155.286) | 25.004 (NA) — Standard deviation was not calculated as only one participant had PK observations. | 532.216 (241.670)
  Day 169 pre-dose: number analyzed (Participants) | 0 | 34 | 0 | 51
  Day 169 pre-dose |  | 50.390 (18.717) |  | 54.031 (30.161)
  Day 169 post-dose: number analyzed (Participants) | 36 | 34 | 51 | 44
  Day 169 post-dose | 469.366 (92.413) | 65.459 (113.805) | 572.071 (200.235) | 57.018 (31.592)
  Day 197: number analyzed (Participants) | 34 | 34 | 52 | 48
  Day 197 | 39.535 (16.655) | 10.808 (9.982) | 39.399 (15.325) | 14.958 (28.728)
  Day 225: number analyzed (Participants) | 37 | 32 | 51 | 49
  Day 225 | 46.885 (21.633) | 1.903 (1.594) | 73.173 (194.836) | 1.979 (1.624)
  Day 253: number analyzed (Participants) | 36 | 33 | 49 | 49
  Day 253 | 45.069 (23.143) | 0.360 (0.343) | 63.950 (77.006) | 0.427 (0.485)
  Day 281: number analyzed (Participants) | 36 | 33 | 49 | 46
  Day 281 | 46.368 (23.349) | 0.086 (0.160) | 54.050 (50.595) | 0.139 (0.340)
  Day 309: number analyzed (Participants) | 33 | 31 | 49 | 46
  Day 309 | 52.409 (23.754) | 0.008 (0.026) | 44.732 (24.888) | 0.018 (0.044)
  Day 365: number analyzed (Participants) | 21 | 22 | 46 | 45
  Day 365 | 2.446 (2.536) | 0 (0) | 1.531 (1.017) | 0.003 (0.014)

ADVERSE EVENTS:
Time Frame: Up to approximately 365 days
Description: Safety Analysis Set: included all participants who received any dose of investigational product.
  All-cause mortality is reported for all randomized subjects in the study.
Groups:
- Population 1: Placebo (Stage I): Participants with SS characterized by moderate to severe systemic disease activity (defined by an ESSDAI score of ≥ 5), were randomized to receive a placebo in Stage I.
- Population 1: VIB4920 (Stage I): Participants with SS characterized by moderate to severe systemic disease activity (defined by a ESSDAI score of ≥ 5), were randomized to receive multiple doses of VIB4920 in Stage I.
- Population 1: VIB4920 (Stage II): Participants with SS characterized by moderate to severe systemic disease activity (defined by an ESSDAI score of ≥ 5), who received VIB4920 in Stage II.
- Population 1: Placebo (Stage II): Participants with SS characterized by moderate to severe systemic disease activity (defined by an ESSDAI score of ≥ 5), who received placebo in Stage II.
- Population 2: Placebo (Stage I): Participants with SS characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), were randomized to receive a placebo in Stage I.
- Population 2: VIB4920 (Stage I): Participants with SS, characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), were randomized to receive multiple doses of VIB4920 in Stage I.
- Population 2: VIB4920 (Stage II): Participants with SS characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), who received VIB4920 in Stage II.
- Population 2: Placebo (Stage II): Participants with SS characterized by moderate to severe subjective symptoms (defined by an ESSPRI score of ≥ 5), and low systemic disease activity (ESSDAI score < 5), who received placebo in Stage II.
Arm/Group | Population 1: Placebo (Stage I) | Population 1: VIB4920 (Stage I) | Population 1: VIB4920 (Stage II) | Population 1: Placebo (Stage II) | Population 2: Placebo (Stage I) | Population 2: VIB4920 (Stage I) | Population 2: VIB4920 (Stage II) | Population 2: Placebo (Stage II)
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/36 | 0/37 | 0/34 | 0/55 | 0/54 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/36 | 1/37 | 3/34 | 1/55 | 3/54 | 1/52 | 2/49
Other Adverse Events (participants affected / at risk) | 18/38 | 20/36 | 24/37 | 22/34 | 21/55 | 21/54 | 20/52 | 21/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Population 1: Placebo (Stage I) (N=38) | Population 1: VIB4920 (Stage I) (N=36) | Population 1: VIB4920 (Stage II) (N=37) | Population 1: Placebo (Stage II) (N=34) | Population 2: Placebo (Stage I) (N=55) | Population 2: VIB4920 (Stage I) (N=54) | Population 2: VIB4920 (Stage II) (N=52) | Population 2: Placebo (Stage II) (N=49)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Population 1: Placebo (Stage I) (N=38) | Population 1: VIB4920 (Stage I) (N=36) | Population 1: VIB4920 (Stage II) (N=37) | Population 1: Placebo (Stage II) (N=34) | Population 2: Placebo (Stage I) (N=55) | Population 2: VIB4920 (Stage I) (N=54) | Population 2: VIB4920 (Stage II) (N=52) | Population 2: Placebo (Stage II) (N=49)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 2 | 4 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 3 | 0 | 3 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 2 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Device allergy (Immune system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 4 | 6 | 6 | 7 | 8 | 9 | 5
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 0 | 5 | 5 | 2 | 6
Oral herpes (Infections and infestations) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 5 | 5 | 4 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 2 | 2 | 0 | 1 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2 | 1 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 4 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 4 | 4 | 2 | 2 | 2 | 4 | 1
Syncope (Nervous system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT04129164/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT04129164/SAP_001.pdf